CLINICAL TRIAL: NCT07054372
Title: Comparison of the Impact of Different Suspension Mediums on ABO Antibody Titres.
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Titres-01
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Healthy Blood Donor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Blood Donor: Healthy Blood Donor
  Interventions: Diagnostic Test: Titres on conventional test tube method with different diluent

INTERVENTIONS:
Diagnostic Test: Titres on conventional test tube method with different diluent — Titres on conventional test tube method with different diluent

SUMMARY:
Accurate estimation of ABO antibody titres is vital in Transfusion Medicine due to their involvement in hemolytic transfusion reactions, hemolytic disease of the fetus and newborn, and solid-organ transplant rejection. Although the conventional tube technique (CTT) remains the gold standard, its standardization is challenging, partly influenced by the choice of diluents. This study aimed to compare commonly used diluents in ABO antibody titration via CTT and analyze the resulting titre variations.

ELIGIBILITY:
Inclusion Criteria:

- Healthy Blood Donor.

Exclusion Criteria:

- Samples from female donors, those with irregular antibodies and reactive to transfusion-transmissible infections on routine testing, were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Blood Donor.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the ABO Antibody Titres. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Dr Meenu Bajpai, MD, Study Director — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided